CLINICAL TRIAL: NCT07130630
Title: Validation and Reliability of the Vietnamese Version of the Pain Self-Efficacy Questionnaire in Patients With Knee Osteoarthritis
Brief Title: Validation and Reliability of the Vietnamese Pain Self-Efficacy Questionnaire in Knee Osteoarthritis
Status: Recruiting | Type: Observational
Sponsor: Khai Quang Nguyen, MD (Other)
Responsible Party: Sponsor-Investigator, Khai Quang Nguyen, MD, Deputy Head, Department of Rehabilitation, Gia Dinh People Hospital
Organization: Gia Dinh People Hospital (Other)
Other Study IDs: 113/NDGĐ- HĐĐĐ
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Knee Osteoarthritis: A single group of patients aged 50+ with clinically diagnosed knee osteoarthritis attending Gia Dinh People's Hospital for outpatient evaluation. Participants will complete the Vietnamese Pain Self-Efficacy Questionnaire (VIET-PSEQ) to assess its psychometric properties.
  Interventions: Other: Completion of Vietnamese Pain Self-Efficacy Questionnaire (PSEQ)

INTERVENTIONS:
Other: Completion of Vietnamese Pain Self-Efficacy Questionnaire (PSEQ) — Participants completed the Vietnamese version of the Pain Self-Efficacy Questionnaire (PSEQ) to assess self-efficacy beliefs related to pain management.

SUMMARY:
This study aims to evaluate the reliability and convergent validity of the Vietnamese version of the Pain Self-Efficacy Questionnaire (VIET-PSEQ) in patients with knee osteoarthritis (KOA). Pain self-efficacy refers to a person's confidence in managing their pain and maintaining daily activities despite it.

A total of 173 patients with KOA will be recruited at Gia Dinh People's Hospital using a convenient sampling method. Eligible participants are 50 years or older, diagnosed with KOA, and experiencing chronic knee pain. They will complete the VIET-PSEQ and other health-related questionnaires during an in-person interview.

The study will assess internal consistency (using Cronbach's alpha), test-retest reliability (by re-assessing a subgroup after 72 hours), and convergent validity by correlating VIET-PSEQ scores with EQ-5D-5L utility index. Additionally, linear regression analysis will examine how age, sex, pain severity, and education level influence pain self-efficacy.

The goal is to determine whether VIET-PSEQ is a reliable and valid tool for measuring pain self-efficacy in Vietnamese patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible for inclusion if they meet all of the following conditions:

* Age ≥ 50 years.
* Diagnosis of knee osteoarthritis (OA) according to the criteria of the American College of Rheumatology (ACR), confirmed by:

  1. application of ACR criteria by the investigator at the time of enrollment; or
  2. a prior diagnosis documented in medical records by a rheumatologist or musculoskeletal specialist.
* Presence of chronic pain related to knee OA, with current pain intensity ≥ 1 on the Visual Analog Scale (VAS).
* No acute flare of knee pain within the past 2 weeks.
* Ability to perform activities of daily living (with or without assistance).
* Ability to read, understand, and complete questionnaires in Vietnamese.
* Willingness to participate and provide informed consent.

Exclusion Criteria:

Participants will be excluded if they meet any of the following conditions:

* Diagnosis of severe psychiatric disorders (e.g., schizophrenia, severe anxiety disorders).
* Presence of cognitive impairment that interferes with the ability to comprehend or answer the questionnaire.
* Diagnosed with systemic inflammatory diseases such as rheumatoid arthritis, systemic lupus erythematosus, or gout.
* Presence of other chronic pain conditions (unrelated to knee OA) that are predominant and significantly affect mobility and daily functioning.
* History of intra-articular injection or knee surgery within the past 3 months.
* Questionnaire (PSEQ) with ≥ 20% of items missing or invalid.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults aged 50 years and older diagnosed with knee osteoarthritis, either newly confirmed at the time of enrollment using the American College of Rheumatology (ACR) criteria or previously diagnosed and documented in the medical records by a specialist. Participants will be recruited from outpatient departments in urban hospitals in Vietnam. The population includes patients with chronic knee pain related to osteoarthritis who are able to perform daily activities and comprehend written Vietnamese.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Internal consistency and test-retest reliability of the Vietnamese version of the Pain Self-Efficacy Questionnaire (VIET-PSEQ) | Baseline and follow-up at Day 3 for test-retest group
  The primary outcomes are the internal consistency and test-retest reliability of the Vietnamese version of the Pain Self-Efficacy Questionnaire (VIET-PSEQ) among patients with knee osteoarthritis. Internal consistency will be assessed using Cronbach's alpha with a threshold of ≥ 0.70. Test-retest reliability will be evaluated using the intraclass correlation coefficient (ICC) calculated from a two-way random-effects model with absolute agreement, based on repeated assessments 3 days apart without clinical intervention.

SECONDARY OUTCOMES:
Convergent validity of the VIET-PSEQ via correlation with EQ-5D-5L index score | At baseline assessment
  To assess the convergent validity of the VIET-PSEQ by analyzing its correlation with the EQ-5D-5L utility index. This aims to explore the association between pain self-efficacy and health-related quality of life in patients with knee osteoarthritis. Correlation will be examined using Spearman's rho or Pearson's r depending on data distribution.

OTHER OUTCOMES:
Regression analysis of predictors of total VIET PSEQ score | At baseline (upon enrollment)
  Linear regression will be conducted to evaluate the association between total VIET PSEQ score and potential predictors including age, gender, pain intensity (VAS), and education level. Assumptions of the linear model will be tested. In case of non-normal distribution, data transformation or alternative models such as quantile regression will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Gia Dinh People's Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results of this study will be shared with other researchers upon reasonable request. The data will be de-identified to protect participant privacy and used solely for academic and non-commercial research purposes.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the primary results. Data will remain accessible for a period of 5 years following this initial release.
Access Criteria: Qualified researchers affiliated with academic institutions or research organizations may access the data by submitting a data use request, including a brief proposal outlining research objectives, methodology, and intended outcomes. Data access is conditional upon signing a data-sharing agreement to ensure ethical use and data protection compliance.